CLINICAL TRIAL: NCT05999240
Title: A Target Engagement Study of Pimavanserin for Behavioral Inflexibility With Open Label Trial for Rigid Rigid-compulsive Behavior in Adolescents and Adults With Autism
Brief Title: Pimavanserin for Rigid-compulsive Symptoms in Autism Spectrum Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: ACADIA Pharmaceuticals Inc. (Industry); University of Kansas Medical Center (Other); Research Foundation for Mental Hygiene, Inc. (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Jeremy Veenstra-vanderweele, MD, New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 8449
Record Dates: First submitted 2023-08-13; First posted 2023-08-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
Keywords: Pimavanserin; Nuplazid; Antiparkinson Agents; Antipsychotic Agents; Serotonin 5-HT2 Receptor Antagonist; Physiological Effects of Drugs; Serotonin Agents; Autism Spectrum Disorder; Autistic Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — pimavanserin

STUDY DESIGN:
Intervention Model Description: This study plans to enroll 30 participants between the ages of 16-40 years old with a diagnosis of autism spectrum disorder to participate in a randomized, placebo-controlled, cross-over designed study. Participants will be randomized to take a single dose of either pimavanserin 34 mg or placebo (Visit 2) three hours before beginning a cognitive neuroscience battery. One week later (Visit 3), participants will take the other medication (placebo or pimavanserin 34 mg) three hours before beginning the cognitive neuroscience battery. After completing the second experimental day, participants will immediately enter the Open Label Trial, where they will take pimavanserin 34 mg for six weeks total, with study visits at 3 weeks (Visit 4) and 6 weeks (Visit 5) to complete safety and primary/secondary outcome measures, followed by a follow-up phone call within 30 days after completing the open label trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Information regarding Masking will be communicated to the investigational pharmacy only - all other staff will remain blind to group assignment throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pimavanserin tartrate (Experimental): Pimavanserin 34 mg white to off-white capsules.
  Interventions: Drug: Pimavanserin Tartrate 34 Mg ORAL CAPSULE [NUPLAZID]
- Placebo (Placebo Comparator): Placebo to Pimavanserin tartrate
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pimavanserin Tartrate 34 Mg ORAL CAPSULE [NUPLAZID] — Participants will be randomized to take a single dose of either pimavanserin 34 mg or placebo at Visit 2.
  Other Names: Nuzplazid
  Arms: Pimavanserin tartrate
Drug: Placebo — Placebo for Pimavanserin Tartrate 34 Mg ORAL CAPSILE [NUPLAZID]
  Arms: Placebo

SUMMARY:
This Phase 2 study examines the safety, tolerability, and preliminary efficacy of pimavanserin in individuals with Autism Spectrum Disorder. Male or female participants aged 16 to 40 years of age will be randomized to receive single doses of either placebo or pimavanserin in this randomized, placebo-controlled, cross-over designed study, followed by open label extension.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn the safety, tolerability and to assess pimavanserin for effects on behavioral rigidity and rigid-compulsive behavior in adolescents and adults with Autism Spectrum Disorder.

Participants who meet protocol criteria will be randomly assigned to receive either pimavanserin or placebo in a 1:1 ratio in the Treatment Period. After completing the second experimental day of the cross-over trial, participants will immediately enter the Open-Label Trial, where they will take pimavanserin 34 mg for six weeks total. There will be 2 recruiting sites with a total sample of 30 participants. Blinding will be maintained by using identical tablets containing either Pimavanserin or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 16 years old and no greater than 40 years old.
* Participants 18 years of age or older or a legally acceptable representative must be able and willing to sign an informed consent document indicating understanding of the protocol and procedures and willingness to participate in full. For adult participants, a parent, caregiver, or other adult informant must also sign an informed consent document indicating understanding the requirements for completing their portion of the study and their willingness to participate. For a participant who is under 18 years of age, a parent or guardian must sign an informed consent document indicating understanding the protocol and procedures and willingness to participate in full. Signed assent indicating understanding and willingness to participate is required of participants under 18 years of age.
* Participant must have a diagnosis of Autism Spectrum Disorder, according to DSM-5 criteria, made by a licensed study psychiatrist or psychologist and supported by the Autism Diagnostic Observation Schedule 2 (ADOS-2) completed at screening or within the past 12 months prior to screening by an appropriately trained professional.
* Participant must have a Clinical Global Impression of Severity for Repetitive Behavior of 4 or greater, as rated by the study psychiatrist or psychologist at Screening and at Baseline
* Participant must have a non-verbal IQ of greater than or equal to 70 as determined by the 4-subtest Wechsler Abbreviated Scale of Intelligence.
* Participant must be able to speak and understand English in order to complete study measures.
* Participant must live with a parent, primary caregiver, or other adult informant who can complete study measures on the basis of spending an average of at least 4 hours per day with the participant
* Parent, primary caregiver, or other adult informant must speak and understand English in order to complete study measures.
* Participant must be able to self-administer study medication or have parent/caregiver be able to administer study medication.
* Participant must be able to swallow study medication whole with liquid.
* Participant or legally acceptable representative must be willing to continue current medication(s) and behavioral intervention(s) and to not add or change medication(s) or behavioral intervention(s) over the full course of the study.

Exclusion Criteria:

* Participant is judged by the Investigator to be unable to perform or comply with all study specific requirements.
* Participant is an employee of an investigator with direct involvement in the proposed study or other studies under the direction of a study investigator, or is a family member of an investigator.
* Participant has a history of any severe or unstable psychiatric condition (e.g., schizophrenia or other psychotic disorder, bipolar disorder, major depressive disorder) that, in the opinion of the Investigator, could confound the interpretation of the study results or put the participant at undue risk. An acute episode of a mood disorder will be considered exclusionary; a participant with a history of mild to moderate mood disorder may be included in the study under the discretion of the Investigator. Other stable psychiatric conditions are permitted at the discretion of the Investigator (e.g., attention deficit hyperactivity disorder, generalized anxiety disorder, etc.).
* Participant has a current or recent history of clinically significant suicidal ideation within the past 6 months, corresponding to a score of 3 or higher (active suicidal ideation with some intent to act, without specific plan) on the Columbia Suicide Severity Rating Scale (C-SSRS), or a history of suicidal behavior within the past year, as validated by the C-SSRS at screening or Day 1.
* Participant has met DSM-5 criteria for a substance abuse disorder within the last 6 months prior to Screening, except for disorders related to caffeine or nicotine.
* Participant has a positive test for an illicit drug or cannabis at Screening or Baseline. Participants who test positive for cannabis and who have a valid prescription may be rescreened if they agree to abstain from the cannabis for the length of their participation in the study. The repeat test must be negative for them to participate in the study.
* Participant is taking a serotonin reuptake inhibitor or antipsychotic medication.
* Participant has had a change to psychotropic medications within the last 2 months
* Participant has received electroconvulsive therapy (ECT) in the last 6 months.
* Participant has received new-onset psychotherapy or has had a change in the intensity of psychotherapy within the 2 months prior to Screening.
* Participant has known allergies, hypersensitivity, or intolerance to Pimavanserin or its excipients.
* Participant has received an investigational drug or used an investigational medical device within 3 months before the planned start of study or is currently enrolled in an investigational study.
* Participant has a body mass index (BMI) <17 or >40 at Screening.
* Participant has a known history of long QT syndrome or family history of sudden death.
* Participant has a history of myocardial infarction, unstable angina, acute coronary syndrome, or cerebrovascular accident (CVA) within the last 4 months. Has greater than NYHA Class 2 congestive heart failure or Class 2 angina pectoris, sustained ventricular tachycardia (VT), ventricular fibrillation, torsade de pointes, or syncope due to an arrhythmia.
* Participant has a history of neuroleptic malignant syndrome/serotonin syndrome.
* Participant has had a seizure within the past 12 months. Individuals with seizure disorders who are on stable seizure medications (i.e., without seizures in the past 12 months) are permitted at the discretion of the Investigator.
* Participant is pregnant or breast-feeding, or planning to become pregnant or breastfeed while enrolled in this study or within 3 months after the last dose of study drug.
* Participant has current evidence, or a history within the previous 3 months prior to screening, of a serious and/or unstable neurologic, cardiovascular, respiratory, gastrointestinal, renal, hepatic, hematologic, or other medical disorder, that, in the opinion of the Investigator, would jeopardize the safe participation of the Participant in the study.
* Participant has a history of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the Investigator, is considered cured with minimal risk of recurrence).
* Participant has a known history of a positive hepatitis C virus (HCV) or human immunodeficiency virus (HIV) test.
* Participant has a Screening or Baseline ECG with a QTcF>450ms when the QRS duration is <120 ms or has a Screening or Baseline ECG with a QTcF>470 ms when the QRS duration is >120 ms.
* Participant has laboratory evidence of hypothyroidism at Screening, as measured by thyroid stimulating hormone (TSH) and reflex free thyroxine (T4). If TSH is abnormal and the reflex free T4 is normal, the Participant may be enrolled.
* Participant has current unstable diabetes or glycosylated hemoglobin (HbAIc) >8% at Screening.
* Participant has other clinically significant laboratory abnormalities that, in the opinion of the Investigator, would jeopardize the safe participation of the study Participant.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact of a single dose of pimavanserin 34 mg versus placebo | Post Intervention, 30 days after study completion
  Assessed using cognitive neuroscience task, comparison between pimavanserin and placebo within participants in single-dose cross-over experiment.
Evaluate pimavanserin for treatment of restricted/repetitive behavior in ASD | 6 weeks of Open-Label treatment
  Assessed using the Repetitive Behavior Scale - Revised (RBS-R) rated at baseline, 3, and 6 weeks. The RBS-R is a 44-item self-report form used to measure the wide range of repetitive behavior in children, adolescents, and adults with Autism Spectrum disorders. The scale consists of six subscales with questions related to Stereotyped Behavior, Self-injurious Behavior, Compulsive Behavior, Routine Behavior, Sameness Behavior, and Restricted Behavior rated between 0 to 3 on severity of each item.

SECONDARY OUTCOMES:
Explore the effects of pimavanserin on an electroencephalogram event-related potential (EEG/ERP) reversal learning test | Post 6-week treatment
  Explore the effects of pimavanserin on an electroencephalogram event-related potential (EEG/ERP) learning task in the cross-over comparison (visits 2 and 3) and again at the end of 6 weeks of open label treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Veenstra-VanderWeele, MD, Principal Investigator — New York State Psychiatric Institute; Matthew Mosconi, PhD, Principal Investigator — University of Kansas Center for Autism Research and Training
Locations (2):
- United States (2):
  - Wakarusa Research Facility, Lawrence, Kansas
  - Center for Autism and the Developing Brain, White Plains, New York

IPD SHARING:
Plan to Share IPD: No